CLINICAL TRIAL: NCT06911385
Title: Augmenting Cerebral Blood Flow Using a Novel Combined Treatment Approach in Patients With Ischemic Stroke: Protocol Development
Brief Title: Augmenting Cerebral Blood Flow in Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00139595; RES0060767 (Other Grant/Funding Number: Health Everywhere: Building an ecosystem of innovation in eHealth and mHealth in Alberta)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Remote ischemic conditioning; Pneumatic Lower limb Compression; Stroke; Cerebral blood flow; Functional near infrared spectroscopy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote ischemic conditioning plus Pneumatic Compression (Experimental)
  Interventions: Device: Arm Remote Ischemic Conditioning plus Pneumatic Compression lower limb

INTERVENTIONS:
Device: Arm Remote Ischemic Conditioning plus Pneumatic Compression lower limb — Arm Remote Ischemic Conditioning (4 cycles) plus Pneumatic Compression lower limb (100 mmHg for 1 hour)

SUMMARY:
The most common type of stroke is ischemic (lack of blood flow to the brain due to a clot blocking a blood vessel). Time is brain and an average of 1.9 million brain nerve cells per minute are destroyed in patients experiencing a typical LVO. The main goal of treatment is to help restore blood flow as quickly as possible and prevent brain tissue and cell death. Acute treatments like clot-busting medication or clot removal by wire are standard of care but are available in comprehensive stroke centers in a few urban centers. Often, patients need to be transferred to these centers via ground or air ambulance, sometimes over hours, and no active treatment can be provided during these transfers.

Enhancing or increasing blood flow to the brain is associated with good outcomes in stroke. This study involves an innovative approach combining two treatment interventions - Remote ischemic conditioning (arms) and Air compression therapy (legs, applied simultaneously to all four limbs, that may help improve blood flow to the brain. Remote Ischemic Conditioning is a type of treatment delivered with the help of a regular blood pressure machine. This does not involve any drug. A typical treatment involves the application of a blood pressure cuff followed by brief sessions of compressions and relaxation on the arm muscles, much akin to blood pressure measurement, but for 5 min. It leads to a transient safe state of less blood flow in arm muscles which initiates the release of molecules and signals transmitted by blood. These signals may then go on to improve blood flow in the brain. Air Compression is delivered by a commercially available device (Normatech Elite). They are inflatable sleeves resembling puffy thigh-high boots that deliver compressive pulses stimulating blood flow in the legs, in a graded manner from the ankles to the thighs. We believe this air compression device may help improve and divert blood flow to stroke-affected areas in the brain.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Both male and female participants will be included
3. History of Stroke Symptoms
4. Baseline modified Rankin scale score < 2
5. Participant or substitute decision-maker able to provide informed consent.

Exclusion Criteria:

1. Injury to the upper arms, lower limbs (from ankles to thighs), or any other musculoskeletal disability/pain that precludes tolerating RIC and/or Pneumatic compression therapy.
2. History of dermatological conditions affecting application of RIC cuff with tissue perfusion sensor and pneumatic compression boots.
3. History of peripheral arterial disease
4. Treatment of ongoing malignancy with expected survival < 6 months
5. Presence of hypertensive urgency and emergency
6. Presence of hemodynamic instability and ongoing pulmonary edema
7. Presence of clinical or imaging signs of raised intracranial, intrathoracic, and /or intra-abdominal pressure.
8. Presence of ongoing systemic infection with antibiotic therapy
9. Pregnant and lactating women
10. Participant not part of other clinical intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention completion | End of intervention at 1 hour
  The primary outcome measure is the feasibility of intervention completion as assessed by proportion of patients able to complete the treatment protocol including pre-treatment assessment, intervention, and post-treatment assessment.

SECONDARY OUTCOMES:
Tolerability of intervention | End of intervention at 1 hour
  The secondary outcome measure is tolerability of intervention as assessed by the 5-point Likert scale (1 Very comfortable, 2 Comfortable, 3 neither comfortable nor uncomfortable, 4 uncomfortable, 5 very uncomfortable).
Change in cortical oxygenation content | End of intervention at 1 hour
  The secondary physiological outcome measure is change in cortical oxygenation content as assessed by continuous wave-fNIRS before and after treatment.
Feasibility of ease of delivery of the intervention | End of intervention at 1 hour
  The secondary feasibility outcome measure is ease of delivery of the intervention individual patients by study team member as assessed by 5-point Likert scale (1-very easy, 2-easy, 3-neither easy nor difficult, 4-difficult and 5-very difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Kate, MD, DM, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after completion of study
Access Criteria: Please contact the principal investigator